CLINICAL TRIAL: NCT06258395
Title: The Effect of Moral Distress on Attitudes Towards Clinical Practice in Nursing Students
Brief Title: Moral Distress in Nursing Students
Status: Completed | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Aysun Acun 3
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-02

CONDITIONS: Moral Distress
Keywords: nurse; nurse education; Moral Distress; Ethics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nursing 2st year: second year nursing students
- Nursing 3st year: third year nursing students
- Nursing 4st year: fourth year nursing students

SUMMARY:
Moral Distress (MD), also known as moral distress, was first defined by Jameton in 1984 as "the distress experienced by a person in situations where it is almost impossible to follow the correct course of action due to institutional constraints, despite knowing the correct action to take." Like all health professionals, nursing students can observe conflicts, ethical dilemmas, ethical and moral problems at the individual, clinical and managerial levels during clinical practice, and can even be directly involved in these problems. This study aimed to investigate the effect of MD on attitudes towards clinical practices in nursing students who have started to provide clinical experience. The study will be conducted with 2nd, 3rd and 4th year students studying in the nursing department of a university.

DETAILED DESCRIPTION:
Competence in the nursing profession is of great importance in quality care practices, nurse leadership in teamwork, academic and clinical performance, both in terms of professionalism and the quality of life of patients. Competence in the profession is possible through clinical practices that allow gaining bedside experience after evidence-based theoretical knowledge. While clinical practices are of great importance for students to gain professional knowledge and skills, they also appear as a cause of stress. Care of the sick individual, not being able to find an adequate guide, lack of a role model, negative relationships with healthcare professionals in the clinic, clinical conditions being inadequate for students' knowledge and skills for practice, fear of making mistakes and failure in students, ethical dilemmas they witness in clinical practices and negative emotions as a result of ethical dilemmas. Many situations such as this increase stress in students. Adding moral distress to students' existing stress sources reduces clinical motivation. In this context, determining nursing students; attitudes towards clinical practices has an important place in improving students; motivation and perceptions of their professional lives. It is impossible to eliminate MD in the nursing profession, which focuses on people and touches people;s quality of life. In this case, it is of great importance to understand MD both in professional life and in nursing education, to agree on precautions and to ensure that students are strengthened in terms of MD. It will also affect the attitudes of students who are successful in MD management towards clinical practices at the desired level, and this will strengthen the quality of life of the individual and the society. This study aimed to investigate the effect of MD on attitudes towards clinical practices in nursing students who have started to provide clinical experience. It is anticipated that the results of this research will contribute to the literature and faculty members who take an active role in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Being a 2nd, 3rd and 4th year student studying in the nursing department.
* Having clinical practice experience.
* Volunteering to participate in the study.

Exclusion Criteria:

* Not volunteering to participate in the study.

Ages: 17 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 2nd, 3rd and 4th year students studying in the nursing department with clinical practice experience.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Moral distress | 05/02/2024-20/02/2024

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Turkey (Türkiye)